CLINICAL TRIAL: NCT06957275
Title: The Effects of Pharyngeal Packing on the Postoperative Gastric Fluid Volume Measured by Ultrasound in Patients Undergoing Functional Endoscopic Nasal Surgery, a Randomized Controlled Double-blinded Non-inferiority Trial
Brief Title: The Effects of Pharyngeal Packing on the Postoperative Gastric Fluid Volume in Patients Undergoing Functional Endoscopic Nasal Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Khaled Abdelfattah Abdallah Sarhan, principal investigator, Asst. professor of anesthesia, Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MD-420-2023
Record Dates: First submitted 2025-04-26; First posted 2025-05-04 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Transanal Endoscopic Surgical Procedures; Residual Volume; Gastric; Ultrasound
Keywords: Ultrasound; Gastric residual volume; Endoscopic sinus surgery

STUDY DESIGN:
Intervention Model Description: In this study, patients undergoing Nasal surgery will be randomized into 2 groups.
  * Group (P): will include the patients who will receive pharyngeal packing
  * Group (C): will include the patients who will not receive pharyngeal packing
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- non packing group (c) (Experimental): will include the patients who will not receive pharyngeal packing
  Interventions: Procedure: Nasal packing
- packing group (P) (Active Comparator): will include the patients who will receive pharyngeal packing
  Interventions: Procedure: Nasal packing

INTERVENTIONS:
Procedure: Nasal packing — group c will not receive pharyngeal packing
  Arms: packing group (P)
Procedure: Nasal packing — Group (P): will include the patients who will receive pharyngeal packing
  Arms: non packing group (c)

SUMMARY:
In this study, the aim is to investigate the effects of Pharyngeal Packing on the perioperative gastric volume in patients undergoing FESS, by ultrasound assessment

DETAILED DESCRIPTION:
Following approval from the Ethics and Research Committee of the anesthesia department, Faculty of Medicine, Cairo University, and obtaining written informed consent from all participating patients meeting the inclusion criteria; patients will be randomly assigned into two groups using a computer-generated random number list with a closed-sealed envelope.

* Group (P): will include the patients who will receive pharyngeal packing
* Group (C): will include the patients who will not receive pharyngeal packing The day before the operation, all patients should be instructed to follow institutional fasting guidelines (a minimum of 2 h for clear fluids, 6 h for a light meal, and 8 h for a meal that included fried or fatty food) On operation day,The patient will attend at the pre-anesthesia room 1 hour before the procedure. A 20 Gauge cannula will be inserted peripherally.

Prophylactic antiemetic (metoclopramide 0.15mg/ kg) will be given slowly intravenously as premedication.

Then a serial ultrasonographic qualitative and quantitative assessment of the gastric antrum of the patients will be done and recorded preoperatively by the anesthetist who will be blinded to the study groups.

A preoperative ultrasonographic examination of the gastric antrum (at the sagittal plane between the left lobe of the liver and pancreas at the level of the aorta) will be performed in the right lateral decubitus position

Ultrasound Assessments:

A standardized scanning technique will be used with a portable sonographic system equipped with a 5- to 2-MHz curved array transducer (GE HealthCare). Subjects will be first placed in the supine position and then in the right lateral decubitus (RLD) position, always in a 45°semirecumbent position. In both of these positions, fluid or semifluid content gravitates preferentially to the antrum, and air or gas is displaced proximally toward the body or fundus, thus facilitating antral sonography (8) During ultrasound imaging, the gastric antrum will be identified in the sagittal to right parasagittal plane using the left lobe of the liver, the pancreas, abdominal aorta, or inferior vena cava as anatomical landmarks. The ultrasonographic assessment will consist of a qualitative and quantitative evaluation of the gastric antrum. The qualitative assessment is aimed at the nature of gastric content (empty, fluid, or solid content). Based exclusively on this qualitative assessment of the antrum, and once the presence of solid content will be ruled out, patients will be classified into 3 grades (12)

* Grade 0 antrum: is defined as the absence of fluid content in both supine and RLD positions, suggesting a "completely empty" state.
* Grade 1 antrum: If fluid content is observed only in the RLD position, but not in the supine position. It correlates with low-volume states compatible with baseline gastric secretions in fasted patients.
* Grade 2 antrum: If fluid is observed in both supine and RLD. The quantitative assessment of the gastric volume will be performed by measuring the cross-sectional area (CSA) of the gastric antrum (antral CSA) between peristaltic contractions, using the free-tracing calibre of the ultrasound unit. This free-tracing method is equivalent to the 2-diameter method of area measurement, and it is simpler and highly reproducible. This validated method allows rapid point-of-care assessment at the bedside, which is relevant for clinical practice (13) Using GE ultrasonography

Then gastric volume will be calculated using the following equation:

Volume (ml) = 27 + 14.6 x Right lateral CSA (cm2

) - 1.28 x age (year) Where Right-lat CSA is the antral CSA measured in the right lateral decubitus. In the operative room, standard monitoring (electrocardiography, pulse oximetry, non-invasive blood pressure, and capnography after intubation) will be applied to the patient.

General Anesthesia (GA) will be induced by another anesthetist who will open the closed envelope and not be blinded to the study groups with intravenous propofol 2 mg/kg, fentanyl 2 mcg/kg, atracurium 0.5 mg/kg, and the trachea will be intubated after mask ventilation for 3 minutes.

Anesthesia will be maintained with IPPV, isoflurane (MAC 1-1.5) in oxygen/air and atracurium 0.1mg/kg as a neuromuscular blocker by the time every 20 minutes. Ventilation will be controlled to maintain an end-tidal CO2 at 30 -35 mmHg.

Following the orotracheal intubation, soft wet pharyngeal packs were placed with gentle maneuvers to avoid damage to the soft palate in patients in group (P). The end of the pharyngeal pack will be hidden inside the mouth of the patient. Patients in both groups were intravenously administered ranitidine (0.5 mg/kg) following the intubation, and ketorolac (30 mg) and pethidine (0.5 mg/kg) at the end of the operation for postoperative analgesia.

Gastric ultrasonographic evaluation will be done at the end of the operation by the same anesthetist who will be blinded to the study group as described before, and the pharyngeal packs of the patients in group(P) will be removed, the residual neuromuscular block will be antagonized with atropine 0.01 m/kg and neostigmine 0.05mg/kg and extubation and suction under vision will be done.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be adult patients (above 18 years), with American Society of Anesthesiologists physical status I-II, scheduled for elective FESS under general anesthesia.

Exclusion Criteria:

* Patients at risk of aspiration (patients with lower esophageal disease such as Hiatus hernia, or GERD and DM).
* Pregnancy.
* Body mass index (BMI) greater than 35 kg/m2.
* Refusal of the patient.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2025-04-26 (Actual); Primary Completion 2025-08-07 (Actual); Study Completion 2025-08-07 (Actual)

PRIMARY OUTCOMES:
The primary outcome of the current study is Gastric residual volume at the end of the procedure. | 4 hours
  The primary outcome of the current study is Gastric residual volume at the end of the procedure.

SECONDARY OUTCOMES:
Quantitative assessment of the risk of aspiration | 6 hours
  Quantitative assessment of the risk of aspiration will be done using three cut-off values for GFV; 1.5 mL/kg, 1.25 mL/kg, and 0.8 mL/kg.
Post operative nausea and vomiting incidence at PACU | 6 hours
  Post operative nausea and vomiting incidence will be assessed at 5-time points using PONV score
Lung ultrasound Score | 6 hours
  Lung ultrasound will be performed before induction of anesthesia and at the end of the operation and using the same curvilinear probe and will be assessed according to the lung ultrasound score
Throat pain at Post anesthesia care unit | 6 hours
  Throat pain will be assessed using VAS

CONTACTS AND LOCATIONS:
Overall Officials: Khaled Sarhan, MD, Principal Investigator — Cairo University
Locations (1):
- Cairo university hospitals, kasralainy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No